CLINICAL TRIAL: NCT06317779
Title: Evaluation of Laparoscopic Cholecystectomy and Concomitant Paraumbilical Hernia Repair
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Mohamed Fazary, Assistant lecturer, Assiut University
Other Study IDs: abdominal laparotomy
Record Dates: First submitted 2024-02-16; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Abdominal Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Umbilical hernia frequently accompanies cholelithiasis. It is possible to repair these hernias after completing cholecystectomy.

DETAILED DESCRIPTION:
Laparoscopy is a type of surgical procedure that allows a surgeon to access the inside of the abdomen and pelvis without having to make large incisions in the skin.

The use of laparoscopy in abdominal surgeries increases for its great benefits over open surgery as:

1)faster recovery, 2)shorter hospital stays 3)decrease blood loss, 4)decreased postoperative pain 5)earlier return to work and resumption of normal daily activity as well as, 6)cosmetic benefits. few studies discuss the efficacy and safety of using Laparoscopy in management of lap cholecyctectomy and concomitant paraumbilical hernia repair

ELIGIBILITY:
Inclusion Criteria:

* Any age, any sex of patients with chronic calcular cholecystitis associated with para-umbilical hernia

Exclusion Criteria:

* Patients with associated diseases such as chronic pulmonary disease, cardiac disease, chronic renal failure.

patients with strangulated para-umbilical hernia

patients with recurrent paraumbilical hernia

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any age, any sex of patients with chronic calcular cholecystitis associated with para-umbilical hernia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Laparoscopic cholecystectomy and concomitant paraumbilical hernia repair | Baseline
  the incidence of recurrence of hernia

SECONDARY OUTCOMES:
Secondary outcomes measures | Baseline
  Decrease duration of operation by doing two by hours minutes operation at same session

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Ali, Study Director — General surgery